CLINICAL TRIAL: NCT03117738
Title: A Phase 1/2, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of AstroStem, Autologous Adipose Tissue Derived Mesenchymal Stem Cells, in Patients With Alzheimer's Disease
Brief Title: A Study to Evaluate the Safety and Efficacy of AstroStem in Treatment of Alzheimer's Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nature Cell Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AST-ADP2-US01
Record Dates: First submitted 2017-04-10; First posted 2017-04-18 (Actual); Results first posted 2021-07-09 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-06

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AstroStem (Experimental)
  Interventions: Drug: AstroStem
- Placebo-Control (Placebo Comparator)
  Interventions: Other: Placebo-Control

INTERVENTIONS:
Drug: AstroStem — Autologous adipose tissue derived mesenchymal stem cells (AdMSC)
  Arms: AstroStem
Other: Placebo-Control — Saline with 30% auto-serum
  Arms: Placebo-Control

SUMMARY:
This is a randomized, double-blind, placebo-controlled, parallel-group comparison study in subjects with Alzheimer's Disease. Following first screening period, subjects will be randomly assigned into one of the following arms: AstroStem and placebo control in a 1:1 ratio. AstroStem or placebo control will be administered via I.V. at Week 0. This procedure will be repeated 9 times at 2-week interval. Subjects will be scheduled for two follow-up visits at Weeks 30 and 52 to evaluate primary and secondary outcome endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 50 and above at the time of signing the Informed Consent form
* Subjects who can understand and provide written informed consent (assent)
* Subjects who have diagnosis of probable mild-to-moderate Alzheimer disease according to NINCDS-ADRDA (National Institute of Neurological and Communicative Disorders and Stroke; Alzheimer's Disease and Related Disorders Association) criteria
* Subjects who have MMSE Score of 16 to 26 at screening
* Subjects who are taking FDA-approved AD medications (donepezil, galantamine, memantine, rivastigmine or their combinations) treatment on a stable dosage for at least 3 months prior to screening.
* Subjects who have one (or more) identified adult caregiver who is able to read, understand, and speak the designated language at the study site; either lives with the subject or sees the subject for ≥2 hours/day ≥4 days/week; and agrees to accompany the subject to each study visit
* Subjects who have a designated study partner who will accompany the subject to all clinic visits and participate in the subject's clinical assessments

Exclusion Criteria:

* Subjects who are females who are pregnant, nursing, or of childbearing potential while not practicing effective contraception
* Subjects who have signs of delirium
* Subjects who have had cortical stroke within the preceding 2 years
* Subjects who have a prolonged QTc interval; >450 msec in male or >470 msec in female at screening
* Subjects who have diagnosis of severe white matter hyperintensity (WMH), which is defined as ≥ 25mm of the deep white matter and ≥ 10mm of the periventricular capping/banding in lengths
* Subjects who have diagnosis of dementia or cause of cognitive impairment other than Alzheimer's disease
* Subjects who have a significant abnormal result in laboratory tests, in the opinion of the investigator
* Subjects who have participated in any investigational drug, stem cell therapy, or device trial within the previous 3 months at screening
* Subjects with any current psychiatric diagnosis other than AD if, in the judgment of the investigator, the psychiatric disorder or symptom is likely to confound interpretation of drug effect, affect cognitive assessments, or affect the subject´s ability to complete the study
* Subjects who are known to have autosomal dominant mutation-associated presenile AD
* Subjects who show signs of AIDS (Acquired Immunodeficiency Syndrome), HBV (Hepatitis B Virus), HCV (Hepatitis C), VDRL (Venereal Disease Research Laboratory)
* Subjects who have any conditions that would contraindicate an MRI, such as the presence metallic objects in the eyes, skin, or heart
* Subjects who have > 4 cerebral microhemorrhages (regardless of their anatomical location or diagnostic characterization as "possible" or "definite"), a single area of superficial siderosis, or evidence of a prior microhemorrhage as assessed by MRI
* Subjects who have history of malignant cancer within the last 5 years (The following is a partial list of conditions that are permissible for study entry: non-metastatic basal and/or squamous cell carcinoma of the skin, in situ cervical, or non-progressive prostate cancer)
* Subjects who have suspected active lung disease based on chest X-ray
* Subjects who are hypersensitive to fetal bovine serum or penicillin
* Subjects who are currently using immunosuppressants, cytotoxic drug, corticosteroids or similar steroidal anti-inflammatory medication (e.g., Prednisone) on a regular basis (exceptions allowed include; regular use of steroidal nasal sprays, topical steroids, and estrogen-replacement therapy)
* Subjects for whom the investigator judges the liposuction can cause any problems
* Subjects who have history of local anesthetic allergy

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-05-09 (Actual); Primary Completion 2019-06-26 (Actual); Study Completion 2019-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - ATP Clinical Research, Costa Mesa, California
  - Syrentis Clinical Research, Santa Ana, California
  - Valden Medical, Honolulu, Hawaii

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- AstroStem: AstroStem: Autologous adipose tissue derived mesenchymal stem cells (AdMSC) 2x10e8 cells
Period: Overall Study
Arm/Group | AstroStem | Placebo-Control
Started | 11 | 10
Completed | 7 | 5
Not Completed | 4 | 5
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Lost to Follow-up | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AstroStem | Placebo-Control | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.4 (7.6) | 75.6 (8.2) | 73.9 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 7 | 5 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not-Hispanic or Latino | 9 | 9 | 18
  White | 10 | 9 | 19
  Black or African American | 0 | 0 | 0
  Asian | 1 | 1 | 2
  American Indian or Alaska Native | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Other | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: cm] | 167.9 (14.4) | 168.3 (9.7) | 168.1 (12.1)
Weight [Mean (Standard Deviation); unit: kg] | 74.8 (17.2) | 64.6 (12.0) | 69.9 (15.5)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 26.3 (4.3) | 22.8 (3.5) | 24.6 (4.3)

OUTCOME MEASURES:

1. Primary Outcome: Treatment Related Adverse Events
Description: Number of subjects with treatment related adverse events as assessed by analysis of adverse events including symptoms, and abnormal findings on physical examination, vital signs, ECG, and standard laboratory examination results
Time Frame: 30 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | AstroStem | Placebo-Control
Number analyzed (Participants) | 11 | 10
Participants | 6 | 3

2. Primary Outcome: ADAS-Cog (Alzheimer's Disease Assessment Scale-cognitive Subscale)
Description: Change of ADAS-Cog (Alzheimer's Disease Assessment Scale-cognitive subscale) from Baseline at Week 30 Score range: 0-70 A score of 70 represents the most severe impairment and 0 represents the least impairment
Time Frame: Baseline and 30 Weeks
Population: 3 of the 11 astrostem groups were dropped out and 1 was violated protocol.
  1 of the 10 Placebo-control groups was dropped out and 2 were violated protocol.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AstroStem | Placebo-Control
Number analyzed (Participants) | 7 | 7
score on a scale | 5.9 (6.8) | 3.0 (5.4)

3. Secondary Outcome: MMSE (Mini-mental Status Examination)
Description: Change of MMSE from baseline at Week 30 Score range: 0-30 A score of 20 to 24 suggests mild dementia, 13 to 20 suggests moderate dementia, and less than 12 indicates severe dementia.
Time Frame: Baseline and 30 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AstroStem | Placebo-Control
Number analyzed (Participants) | 7 | 7
score on a scale | -3.4 (2.8) | -1.4 (2.8)

4. Secondary Outcome: CDR-SOB (Clinical Dementia Rating-Sum of Boxes)
Description: Changes of CDR-SOB from baseline at Week 30 Score range: 0-18.0 0 = normal, 0.5-4.0 = questionable cognitive dementia, 4.5-9.0 = mild dementia, 9.5-15.5 = moderate dementia, and 16.0-18.0 = severe dementia
Time Frame: Baseline and 30 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AstroStem | Placebo-Control
Number analyzed (Participants) | 7 | 7
score on a scale | 1.3 (1.7) | 0.9 (1.5)

5. Secondary Outcome: NPI (Neuropsychiatric Inventory)
Description: Changes of NPI from baseline at Week 30 Score range: 0-144 higher score indicates higher disturbance.
Time Frame: Baseline and 30 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AstroStem | Placebo-Control
Number analyzed (Participants) | 7 | 7
score on a scale | -1.4 (8.5) | -5.7 (11.5)

6. Secondary Outcome: GDS (Geriatric Depression Scale)
Description: Changes of GDS from baseline at Week 30 Score range: 0-15 Scores of 0-4 are considered normal, depending on age, education, and complaints; 5-8 indicate mild depression; 9-11 indicate moderate depression; and 12-15 indicate severe depression.
Time Frame: Baseline and 30 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AstroStem | Placebo-Control
Number analyzed (Participants) | 7 | 7
score on a scale | -0.3 (1.3) | 0.3 (2.1)

7. Secondary Outcome: ADCS-ADL (Alzheimer's Disease Cooperative Study Activities of Daily Living)
Description: Change of ADCS-ADL from baseline at Week 30 Score range: 0-78 Lower score indicates greater severity.
Time Frame: Baseline and 30 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AstroStem | Placebo-Control
Number analyzed (Participants) | 7 | 7
score on a scale | -4.4 (9.0) | -4.7 (9.8)

8. Secondary Outcome: C-SSRS (Columbia Suicide Severity Rating Scale)
Description: Changes of C-SSRS from baseline at Week 30 Score range: 0-25 Higher score indicates higher severity.
Time Frame: Baseline and 30 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AstroStem | Placebo-Control
Number analyzed (Participants) | 11 | 10
score on a scale | -2.1 (6.6) | 0.0 (0.0)

ADVERSE EVENTS:
Time Frame: 52 weeks
Arm/Group | AstroStem | Placebo-Control
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 3/11 | 1/10
Other Adverse Events (participants affected / at risk) | 3/11 | 2/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AstroStem (N=11) | Placebo-Control (N=10)
oesophageal squamous cell carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute Pulmonary Oedema (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AstroStem (N=11) | Placebo-Control (N=10)
Open Angle Glaucoma (Eye disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Reflux Disease (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Infusion Site Reaction (General disorders) | 1 | 0
Oedema Peripheral (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Abnormal Loss of Weight (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Agitation (Psychiatric disorders) | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Study Protocol (2019-03-04): https://cdn.clinicaltrials.gov/large-docs/38/NCT03117738/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-10): https://cdn.clinicaltrials.gov/large-docs/38/NCT03117738/SAP_001.pdf
  • Informed Consent Form (2017-06-26): https://cdn.clinicaltrials.gov/large-docs/38/NCT03117738/ICF_002.pdf